CLINICAL TRIAL: NCT02118740
Title: Bone Marrow Collection in Healthy Volunteers
Brief Title: Bone Marrow Collection in Healthy Volunteers (iCell)
Acronym: iCell
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amarna Stem Cells BV (Industry)
Collaborators: Neuroplast (Industry)
Responsible Party: Sponsor
Other Study IDs: NL44976.068.13; A2013SCI-01 (Other: Sponsor Identification number)
Record Dates: First submitted 2014-03-18; First posted 2014-04-21 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Cord Injury
Keywords: Autologous Stem Cells; Spinal Cord Injury; Preclinical
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — A stem cell specimen will be retained to enable verification in the future
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a observational study in which healthy found volunteers are recruited to donate 50 ml of bone marrow aspirate to enable preclinical studies to obtain proof of concept and safety of a bone marrow derived stem cell preparation named AMARCELL. The prepared AMARCELL is only for animal studies and after completion of the preclinical program, the intention of AMARCELL is to treat humans with a traumatic Spinal cord injury.

DETAILED DESCRIPTION:
Coded anonymized patient data

ELIGIBILITY:
Inclusion Criteria:

* Men in the age range of 21-30 years and/or women in the age range of 21-30 years and taking birth control medication to prevent pregnancy
* Written informed consent
* Healthy as concluded by the answers given to questions in a short health questionnaire

Exclusion Criteria:

* Pregnancy or lactation period
* Volunteers who are unable to comply with the rules of this project. Important is if the volunteer can not follow the schedule of the appointments.
* Abuse of alcohol, medicines or illicit drugs.
* Legally protected people

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-12-30 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of mononuclear cells include hematopoietic stem and progenitor cells in AMARCELL | 3 days
  Important is to have more than 2 million mononuclear cells (MNCs) include hematopoietic stem and progenitor cells in the end product AMARCELL

SECONDARY OUTCOMES:
Absence of contamination with infectious agents especially bacteria and pseudomonas | 3 days
  The end product has to be sterile and will be tested for contamination. No culture after plating on growth medium (after 14 days) and no foreign non-human particles in the sample using Polymerase Chain Reaction techniques (after 6 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Harry Steinbusch, Prof.dr., Study Director — University Maastricht; Gerard Bos, Prof.dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The bone marrow characteristics shall be published as part of the preclinical studies and in particular as a request of the METC